CLINICAL TRIAL: NCT00189683
Title: Xeloda Vs Monitoring in Advanced Colorectal Cancer Responsive to Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Européenne de Recherche en Oncologie (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AERO-MC04
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Procedure: Monitoring
Procedure: Xeloda

SUMMARY:
To compare maintenance chemotherapy with Xeloda to control after best response with first line chemotherapy in advanced colorectal cancer. Main endpoint is progression free survival. A total of 300 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic colorectal cancer (confirmed histologically) with objective response or stabilization after at least 6 cycles of first line chemotherapy (treatment of choice is selected freely by the investigator according to the recommendations and consensus in force),
* The interval between completion of first line chemotherapy and randomization should not exceed 4 weeks
* Age>18 years
* ECOG status 0 to 2
* Biological criteria prior to any chemotherapy:

Neutrophils>1.5 109 g/l, platelets>100 109/l, haemoglobin>10 g/dl, Creatininaemia<150 mol/l, bilirubinaemia<2x normal level

* Signed informed consent
* Life expectancy > 3 months

Exclusion Criteria:

* Metastatic colorectal cancer treated with more than one modality of first line chemotherapy (including oral fluoropyrimidines)
* Tumour progression after first line chemotherapy or before randomization
* Other tumour pathology
* Symptomatic cerebral metastases
* Any severe uncontrolled disease in addition to colorectal cancer (in particular decompensated cardiac failure (LVEF<50%) or coronary insufficiency)
* Lack of integrity of the upper GI tract: malabsorption syndrome or major surgery of the stomach or the small intestine
* Severe renal impairment (creatinine clearance < 30 ml/min)
* Severe psychiatric disorder (other than controlled depressive syndrome)
* Patient participating in another experiment
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fabre-Guillevin, MD, Principal Investigator — AERO; Eric Van Cutsem, MD, Principal Investigator — BGDO; Marc Polus, MD, Principal Investigator — BGDO
Locations (1):
- AERO, Créteil, France